CLINICAL TRIAL: NCT00717431
Title: Medical vs Electrical Therapy for Temporal Lobe Epilepsy
Brief Title: A Multicenter Study of Hippocampal Electrical Stimulation (HS, in Mesial Temporal Lobe Epilepsy
Acronym: METTLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrolment
Sponsor: University of Calgary (Other)
Collaborators: University of Western Ontario, Canada (Other); University of Toronto (Other); Dalhousie University (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Dr. Sam Wiebe, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20492
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Temporal Lobe Epilepsy
Keywords: Deep Brain Stimulation; Seizures; Epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Seizures; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hippocampal Stimulation (Experimental): Hippocampal Stimulation (Stimulator is turned ON) Surgical Intervention
  Interventions: Procedure: Hippocampal Electrical Stimulation
- Hippocampal Implantation (Sham Comparator): Hippocampal Implantation (Stimulator is turned OFF)Surgical Intervention
  Interventions: Procedure: Hippocampal Electrical Stimulation

INTERVENTIONS:
Procedure: Hippocampal Electrical Stimulation — Surgical Implantation of electrode and stimulator

SUMMARY:
The primary goal is to determine whether hippocampal electrical stimulation (HS) is safe and more effective than simply implanting an electrode in the hippocampus without electrical stimulation (HI), in patients with mesial temporal lobe epilepsy (MTLE). This will be assessed by the rate of complex partial seizures per person-month over 6 months of follow-up in HS vs. HI. There are two treatment arms: 1) Hippocampal Electrode Implantation with Stimulation (HS). 2) Hippocampal Electrode Implantation without stimulation (HI). The investigators expect to demonstrate that HS is safe and superior to HI in controlling seizures in patients with MTLE.

DETAILED DESCRIPTION:
This is a multicentre, parallel-group, double blind randomized controlled trial involving patients with MTLE who may be candidates for resective surgery or whose memory function precludes resective surgery. Eligible patients will be randomized in a 2:1 ratio into hippocampal electrode implantation with stimulation (HS), or hippocampal electrode implantation without stimulation (HI). Patients will be followed for seven months after randomization. One month will be devoted to adjustment of interventions, and 6 months to follow-up and outcome assessment. At the end of seven months, all patients will be offered the option of HS, electrode removal, surgical therapy or medical therapy, based on best evidence and patient preference.

Primary Question: In patients with MTLE, over a 6-month period:

Is continuous HS plus medical therapy (MT) more efficacious than hippocampal implantation (HI) plus MT in reducing seizure frequency?

Secondary Questions: In patients with MTLE, over a 6-month period:

1. Is HS safe?
2. What is the effect of HS on cognition, mood, and quality of life?
3. What is the effect of HS on psychiatric morbidity?
4. Is the efficacy of HS associated with the presence, location and amount of interictal hippocampal spikes on depth electrode recordings?

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or Bilateral Mesial Temporal lobe Epilepsy.
* Age ≥ 18 years.
* Global IQ ≥70.
* Failure of ≥ 2 AEDs approved for treatment of partial seizures, used alone or in combination at recommended dosages.
* Average ≥ 3 seizure-days per month in prior 6 months during which disabling seizures occurred. Disabling seizures are defined as complex partial seizures with or without secondary generalization, or as simple partial seizures that are noticeable by others or interfere with function.
* Ability to complete self-administered questionnaires.
* Availability of reliable collateral historian or witness.
* Patient preference for non-resective surgery, or not a candidate for mesial temporal resection.
* Give written informed consent.

Exclusion Criteria:

* Extratemporal or multifocal epilepsy.
* MRI evidence of potentially epileptogenic lesions outside the mesial temporal region.
* Lesions precluding electrode implantation (eg, vascular malformations, vascular tumors).
* Severe hippocampal sclerosis that in the surgeon's opinion precludes accurate electrode placement.
* Brain lesions that demand prompt surgical therapy (eg, malignant tumors, vascular malformations).
* Progressive neurological disorders (eg, malignant tumor, dementia, degenerative disorders).
* Medical or psychiatric conditions precluding surgery or interfering with adherence to treatment and follow-up.
* Planned pregnancy during the study. Women of child-bearing age will require a negative pregnancy test and adequate contraception methods.
* Ongoing or planned participation in other studies of new epilepsy therapies.
* Contraindication for stereotactic surgery, e.g. bleeding diathesis, anticoagulants, treatment with valproate at the time of surgery (risk of bleeding).
* Any condition that would make participation in the trial detrimental to the patient's health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rate of complex partial seizures (with or without secondary generalization) per person-month over 6 months of follow-up. | Months 1-7

SECONDARY OUTCOMES:
Cognitive function: Change in mean scores from baseline to end of study. | Months 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wiebe, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Clinical Neurosciences, Calgary, Alberta, Canada